CLINICAL TRIAL: NCT02803333
Title: Symptoms, Toxicity Prevalence and Quality of Life Benefit of Targeted Therapies and Immunotherapies in Lung Cancer Patients: An Observational Prospective Cohort Study Within the Total Cancer Care Population
Brief Title: Oncology Research Information Exchange Network (ORIEN) Lung Cancer Study
Acronym: ORIEN
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: PatientsLikeMe (Other); Ohio State University Comprehensive Cancer Center (Other); AstraZeneca (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-18515
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: NSCLC; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Thoracic Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Thoracic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data Capture Participants: This is a prospective observational cohort study of advanced non-small cell lung cancer patients (stage 3b/4) receiving treatment at the Moffitt Cancer Center (MCC) or The Ohio State Comprehensive Cancer Center (OSUCCC) to assess treatment impact at monthly intervals from baseline to 6 months post-enrollment.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
The Moffitt Cancer Center and PatientsLikeMe.com (PLM), an online patient community, are working together to better understand the patient's entire lung cancer experience, both inside and outside the doctor's office. By combining the data that is captured by their care team in the clinic with the data participants enter at their home on PatientsLikeMe.com, the investigators hope to improve patient-physician treatment decisions, so that the patient's personal treatment goals and quality of life have the highest chances of being fulfilled.

DETAILED DESCRIPTION:
The aim of the study is to assess the real-world patient experience by evaluating the patients' quality of life, treatment toxicities, and clinical measures over a 6-month period. The ultimate goal of this research is to improve patient-physician treatment decisions, so that the patient's personal treatment goals and quality of life have the highest chances of being fulfilled.

Aim 1. To track the toxicities/side-effects of FDA approved molecular targeted agents, immunotherapies, and combinations of treatments for NSCLC in a clinical setting for six months.

Aim 2. To assess the impact of these treatment regimens on patient toxicities, symptoms, function, and quality of life, after adjustment for clinical factors and patient characteristics during the 6 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Diagnosed with metastatic (stage 3b/4) non-small cell lung cancer (NSCLC)
* The total combined sample size must include at least 100 people who received one or more treatments of PD-1/PDL-1 inhibitor treatment (immunotherapy), and 50 patients who received an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI). Patients receiving any other treatments will be tracked for treatment outcomes, as well as to serve as comparison participants during data analyses of outcomes associated with PD-1/PDL-1 or EGFR-TKI).
* Consented separately to the Total Cancer Care (TCC) protocol
* Have access to the internet
* Willing to enroll in the free online health tracking and patient community "PatientsLikeMe"

Exclusion Criteria:

* Patients enrolled in Phase I clinical trial protocols
* Patients enrolled in Phase II, III or IV clinical trials involving blinded therapies (patients in open label trials will be eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced non-small cell lung cancer patients (stage 3b/4) receiving treatment at the Moffitt Cancer Center (MCC) or The Ohio State University Comprehensive Cancer Center (OSUCCC)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Cancer Treatment Changes | 6 months post enrollment
  Clinical, molecular, and patient-reported data will be collected from participants. Participants will be asked if their treatment course has changed and, if so, what changes have occurred. These questions are primarily meant to identify the number of patients who were switched from one treatment regimen (e.g., chemotherapy) to either PD-1/PDL-1 inhibitor treatment (immunotherapy) or tyrosine kinase inhibitors (TKIs).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Schabath, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/